CLINICAL TRIAL: NCT06767007
Title: Evaluation of the Efficiency and Safety of Stereotactic Body Radiation Therapy Combined With PD-1 Antibody in the Treatment of Unresectable Locally Recurrent Rectal Cancer: A Prospective, Multicenter, Single-Arm, Open Label, Phase II Study
Brief Title: SBRT + PD-1 Antibody in Unresectable Locally Recurrent Rectal Cancer（SPARKLE）
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Fudan University (Other); Sun Yat-sen University (Other); Yunnan Cancer Hospital (Other); Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Huang, Deputy director of the colorectal surgery, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2024300
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Unresectable Locally Recurrent Rectal Cancer
Keywords: Unresectable Locally Recurrent Rectal Cancer; Stereotactic Body Radiation Therapy; PD-1 monoclonal antibody
MeSH Terms: interventions — Radiosurgery; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT+PD1 (Experimental): Participants of experimental arm (SBRT+PD-1 monotherapy group) will receive following treatments by sequences: Chemotherapy combined with PD-1 therapy for 1 cycle → SBRT treatment → Chemotherapy combined with PD-1 therapy for 3-6 cycles (assessment 6 weeks after SBRT treatment) → Surgery/Maintenance therapy.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Drug: PD1; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Patients will begin SBRT treatment within 2 weeks after the first round of chemotherapy. Intensity-modulated radiation therapy (IMRT) technology will be used, with a target gross tumor volume (GTV) of 5-8Gy/5 sessions, a total dose of 25-40Gy equivalent to a biological effective dose (BED) of 37.5-72Gy, administered from Monday to Friday. For patients who have previously received pelvic radiotherapy, the re-irradiation dose will be 3-5Gy/5 sessions, a total dose of 15-25Gy equivalent to a BED of 19.5-37.5Gy, administered from Monday to Friday.
Drug: PD1 — The PD-1 monoclonal antibody used is Sintilimab 200mg every 3 weeks
Drug: Chemotherapy — First-line chemotherapy regimen of rectal cancer, using a second-line regimen primarily based on fluorouracil, such as a tri-weekly CAPOX or a bi-weekly mFOLFOX6/FOLFIRI/FOLFOXIRI + targeted therapy

SUMMARY:
This is a prospective study to delve into the therapeutic benefits of combining stereotactic body radiation therapy (SBRT) with PD-1 monoclonal antibody treatment for patients with unresectable locally recurrent rectal cancer (ULRRC). Our aim is to ascertain the safety of this approach and to offer robust, evidence-based medical guidance for the management of ULRRC using this innovative combination therapy.

Researchers will combine SBRT with PD-1 for ULRRC to see if this treatment can provide a benefit of survival.

Participants will:

1. Receive chemotherapy combined with PD-1 therapy for 1 cycle → SBRT treatment → Chemotherapy combined with PD-1 therapy for 3-6 cycles (assessment 6 weeks after SBRT treatment) → Surgery/Maintenance therapy.
2. Visit the clinic once every 3 months for checkups and tests

DETAILED DESCRIPTION:
This clinical trial is a prospective, open-label, Phase II study. Patients with unresectable locally recurrent rectal cancer(ULRRC) by the multidisciplinary team (MDT) , and where the radiation oncology department within the MDT does not consider the presence of organs at risk (OARs) to affect the execution of SBRT, and who may benefit from improved progression-free survival or the creation of an R0 resection opportunity, are eligible for enrollment. Enrolled patients will receive high-dose fractionated radiotherapy of 5-8Gy per session, for a total of 5 sessions, with chemotherapy based on 5-FU before and after radiotherapy. Imaging assessments for surgical feasibility will be conducted 6 weeks (±2 weeks) after radiotherapy, and the MDT will decide on radical surgery, maintenance chemotherapy, or withdrawal 8 weeks (±2 weeks) after radiotherapy.

Participants will receive:

1 cycle of chemotherapy combined with PD-1 therapy → SBRT treatment → 3-6 cycles of chemotherapy combined with PD-1 therapy (assessed 6 weeks after SBRT treatment) → Surgery/Maintenance therapy.

Protocol of Stereotactic Body Radiation Therapy (SBRT):

Patients will begin SBRT treatment within 2 weeks after the first round of chemotherapy. Intensity-modulated radiation therapy (IMRT) technology will be used, with a target gross tumor volume (GTV) of 5-8Gy/5 sessions, a total dose of 25-40Gy equivalent to a biological effective dose (BED) of 37.5-72Gy, administered from Monday to Friday. For patients who have previously received pelvic radiotherapy, the re-irradiation dose will be 3-5Gy/5 sessions, a total dose of 15-25Gy equivalent to a BED of 19.5-37.5Gy, administered from Monday to Friday.

Protocol of PD-1 Monoclonal Antibody:

The PD-1 monoclonal antibody used is Sintilimab 200mg, administered intravenously on the first day.The study requires completion of at least 4 cycles of PD-1 monotherapy before and after SBRT to be considered eligible.

Protocol of Chemotherapy Regimen:

The choice of chemotherapy drugs will be at the discretion of the physician, based on the first-line chemotherapy regimen, using a second-line regimen primarily based on fluorouracil, such as a tri-weekly CAPOX or a bi-weekly mFOLFOX6/FOLFIRI/FOLFOXIRI + targeted therapy. Best supportive care will be provided during chemotherapy or chemoradiation.

Six weeks (±2 weeks) after the completion of high-dose fractionated radiotherapy, the MDT will assess patients through enhanced CT scans and pelvic MRI to determine disease resectability. If feasible, surgery will be performed 8 weeks (±2 weeks) after chemoradiation. The specific surgical approach depends on the location of recurrence and adjacent structures, as determined by the surgeon. Postoperative adjuvant chemotherapy will be administered based on the assessment by the MDT; if surgery is not possible, maintenance chemotherapy or withdrawal will be considered.

Patients who have completed the treatment or those who have not completed the treatment due to intolerable toxic reactions but have not shown tumor progression will be followed up every 3 months. The follow-up will include physical examinations, CT scans (every 3-6 months), pelvic MRI (3 months, 6 months, and the first year after SBRT treatment, then every 6-12 months thereafter), and colonoscopy examinations (once a year during the first, third, and fifth years of treatment). For patients who have already shown tumor progression, telephone follow-ups will be conducted every 3 months until death. During the follow-up, information on subsequent antitumor treatments and survival data of the patients will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Before implementing procedures related to the research protocol rather than routine care, informed consent forms with the subject's voluntary signature and dated must be obtained in accordance with regulations and institutional guidelines;
2. Patients with pMMR/MSS colorectal cancer;
3. Age between 18 and 75 years;
4. Tumor recurrence confirmed by histology, cytology, or imaging, and the multidisciplinary team (MDT) including surgeons assesses that the recurrent lesion cannot achieve a one-stage R0 resection (unresectable is defined as: 1. Pelvic MRI showing sacral infiltration at or above S2, 2. And/or lateral pelvic wall invasion, 3. And/or obturator vascular nerve infiltration, 4. After MDT discussion, there are no indications for a one-stage R0 resection, 5. The patient refuses total pelvic exenteration or debulking surgery);
5. Locally recurrent rectal adenocarcinoma without clear distant metastasis at diagnosis/MDT team assesses oligometastases as resectable/controllable (UICC 8th edition);
6. No prior radiotherapy, or a gap of more than 6 months between the completion of initial radiotherapy and the start of retreatment, with a previous radiotherapy dose of less than 50.4Gy, and no late toxicity in the small bowel or bladder;
7. ECOG performance status 0-1;
8. Peripheral blood counts and liver and kidney functions within the following allowed ranges (tested within 15 days before treatment start):

   * White blood cells (WBC) ≥ 3.0×10^9/L or Absolute Neutrophil Count (ANC) ≥ 1.5×10^9/L;

     * Hemoglobin (HGB) ≥ 80 g/L;

       * Platelets (PLT) ≥ 100×10^9/L;

         * Liver transaminases (AST/ALT) < 3.0 times the upper limit of the normal range;

           * Total bilirubin (TBIL) < 1.5 times the upper limit of the normal range;

             * Creatinine (CREAT) < 1.5 times the upper limit of the normal range;
9. No history of other malignancies, not pregnant or breastfeeding, and should use effective contraception during the study period and for 6 months after the last administration;
10. Expected survival ≥ 12 months.

Exclusion Criteria:

1. Patients with a history of severe drug allergies (including allergies to platinum-based agents, 5-FU, LV, and 5-HT3 receptor antagonists);
2. Patients who have participated in or are currently participating in other clinical trials within 4 weeks of enrollment;
3. History of receiving anti-PD-1, PD-L1, PD-L2, CTLA-4, or any other specific T-cell co-stimulation or checkpoint pathway targeted therapies;
4. Severe electrolyte abnormalities;
5. Presence of gastrointestinal diseases, such as active ulcers of the stomach or duodenum, ulcerative colitis, or unresected tumors with active bleeding; or other conditions that may lead to gastrointestinal bleeding or perforation; or gastrointestinal perforations that have not healed after surgical treatment;
6. History of arterial thrombosis or deep vein thrombosis within 6 months; history of bleeding or evidence of bleeding tendency within 2 months;
7. Pregnant or breastfeeding women or women who may become pregnant with a positive pregnancy test before the first dose; or female participants who are unwilling to strictly use contraception during the study period and their partners;
8. Brain metastases with a diameter greater than 3cm or a total volume greater than 30cc;
9. Clinical or radiological evidence of spinal cord compression, or tumors within 3 millimeters of the spinal cord on MRI;
10. History or concurrent presence of other active malignant tumors (except for malignant tumors that have been treated curatively and have not recurred for more than 3 years or carcinoma in situ that can be cured with adequate treatment);
11. Combined with severe electrocardiogram abnormalities or active coronary artery disease within 12 months before participating in the study, severe/unstable angina or newly diagnosed angina or myocardial infarction, New York Heart Association (NYHA) Class II or higher congestive heart failure;
12. Patients with active infections (infections causing fever above 38°C);
13. Patients with poorly controlled hypercalcemia, hypertension, diabetes;
14. Patients with severe pulmonary diseases (interstitial pneumonia, pulmonary fibrosis, severe emphysema, etc.);
15. Patients with mental disorders affecting clinical treatment or a history of central nervous system diseases;
16. Patients with severe complications (intestinal obstruction, renal insufficiency, liver dysfunction, cerebrovascular disorders, etc.);
17. Any toxicity of grade 2 or above from previous treatments that has not yet resolved (except for anemia, alopecia, and skin pigmentation);
18. Any medical condition that is unstable or would affect patient safety and compliance with the study;
19. Patients deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
1 year PFS | 1 year
  1 year Progression-Free Survival Rate

SECONDARY OUTCOMES:
1 year OS | 1 year
  1 year Overall Survival Rate
ORR | 1 year
  Overall Response Rate
DCR | 1 year
  Disease Control Rate
R0 resection rate | 1 year
  R0 resection rate in participants
2 years PFS | 2 years
  2 years Local Progression-Free Survival Rate
2 years OS | 2 years
  2 years Overall Survival Rate
Acute Toxic Reaction | 1 year
  Acute Toxic Reaction of SBRT and PD-1 Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jun Huang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No